CLINICAL TRIAL: NCT00003923
Title: Phase II Study of Photodynamic Therapy With PHOTOFRIN (Porfimer Sodium) for Injection in Patients With Malignant Bile Duct Obstruction
Brief Title: Photodynamic Therapy in Treating Patients With Cancer of the Bile Duct, Gallbladder, or Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-015; P30CA008748 (NIH); MSKCC-99015; NCI-G99-1525
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer; Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; cholangiocarcinoma of the gallbladder; cholangiocarcinoma of the extrahepatic bile duct; adult primary cholangiocellular carcinoma
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Pancreatic Neoplasms | interventions — Dihematoporphyrin Ether

INTERVENTIONS:
Drug: porfimer sodium

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. This may be effective treatment for cancer of the bile duct, gallbladder, or pancreas.

PURPOSE: Phase II trial to determine the effectiveness of photodynamic therapy in treating patients who have cancer of the bile duct, gallbladder, or pancreas.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and efficacy of photodynamic therapy using porfimer sodium in patients with unresectable malignant bile duct obstruction.

OUTLINE: Patients are stratified according to tumor location (proximal vs distal). Patients receive porfimer sodium IV over 3-5 minutes on day 1, followed by percutaneous or endoscopic laser light treatment on day 3. Patients achieving partial response or complete response accompanied by an increase in total bilirubin or cholangitis may repeat treatment for a maximum of 3 courses. Patients are followed weekly for 1 month, and then monthly for 1 year.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven malignant bile duct obstruction with obstructive jaundice Primary carcinoma of bile duct, gallbladder, or pancreas OR Metastatic bile duct disease Successful insertion of a percutaneous drain or endoscopic stent Unresectable disease OR Resectable disease but refusal of surgery Prior biliary plastic or metallic stent allowed, if requiring stent replacement due to recurrent jaundice or routine plastic stent change No erosion of biliary tumors into major blood vessels No evidence of bile duct perforation

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin at least 2 mg/dL Renal: Not specified Other: No history of allergies or hypersensitivity to porphyrins No porphyria No cholangitis or pancreatitis

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy or brachytherapy to the abdomen Surgery: See Disease Characteristics Other: No other prior or concurrent experimental or investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 1999-03; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gerdes, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States